CLINICAL TRIAL: NCT02762487
Title: RELIEF Europe Study. A Prospective, Multicenter Study of RefluxManagement With the LINX® System for Gastroesophageal Reflux Disease After Laparoscopic Sleeve Gastrectomy
Brief Title: RELIEF Europe Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Torax Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4700
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: GERD; Gastroesophageal Reflux Disease; Obesity; LSG; Laparoscopic Sleeve Gastrectomy
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LINX arm (Experimental): Previous LSG patient will be treated with the LINX device and serve as their own control
  Interventions: Device: The LINX® Reflux Management System

INTERVENTIONS:
Device: The LINX® Reflux Management System — The LINX device is a permanent implant placed at the area of the lower esophageal sphincter (LES) and is designed to augment a weak LES and minimize or eliminate GERD-related symptoms.
  Other Names: LINX device

SUMMARY:
The purpose of this study is to evaluate the LINX device in patients who have previously undergone laparoscopic sleeve gastrectomy (LSG) for obesity and have chronic gastroesophageal reflux disease (GERD). The study will monitor safety and changes in reflux symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic sleeve gastrectomy (LSG) for obesity >12 months prior to proposed device implantation date.
* Patient is a surgical candidate, i.e. is able to undergo general anesthesia and laparoscopic surgery.
* Documented pathologic esophageal acid exposure by pH monitoring per institution's standard of care (i.e. total distal ambulatory esophageal pH< 4 for ≥ 5.3% (BRAVO) or ≥4.5% (transnasal) or abnormal DeMeester Score (>14.72) within 12 months of proposed implantation date (After Sleeve Gastrectomy).

NOTE: SUBJECTS SHALL HAVE DISCONTINUED ALL GERD MEDICATIONS FOR AT LEAST 7 DAYS PRIOR TO TESTING WITH THE EXCEPTION OF ANTACIDS, WHICH MAY BE TAKEN UP UNTIL THE MORNING OF THE VISIT.

* Chronic GERD symptoms despite maximum medical therapy for the treatment of reflux.
* Age ≥ 21 years
* At least 30% loss of excess weight from date of original LSG surgery.
* Patient is willing and able to cooperate with follow-up examinations.
* Patient has been informed of the study procedures and the treatment and has signed an informed consent form.

Exclusion Criteria:

* Suspected or known allergies to titanium, stainless steel, nickel, or ferrous materials.
* Prior surgery in the area of the gastroesophageal junction (GEJ), including prior hiatal hernia repair.
* Presence of ˃3 cm hiatal hernia as determined by endoscopy or barium esophagram.
* Subject had any major complications related to the laparoscopic sleeve gastrectomy that may interfere with, or increase the risks of the LINX procedure (such as, but not limited to, leaks from the gastric remnant and infection at the sleeve gastrectomy).
* Plans to surgically revise the gastric pouch (either known preoperatively or decided intraoperatively).
* Currently being treated with another investigational drug or investigational device.
* Suspected or confirmed esophageal or gastric cancer or prior gastric or esophageal surgery or endoscopic intervention for GERD (with the exception of sleeve gastrectomy).
* Distal amplitude <35 mmHg or <70% peristaltic sequences.
* Presence of esophagitis - Grade C or D (LA Classification). BMI >35.
* Symptoms of dysphagia more than once per week within the last 3 months.
* Diagnosed with Scleroderma.
* Diagnosed with an esophageal motility disorder such as but not limited to achalasia, nutcracker esophagus, or diffuse esophageal spasm or hypertensive LES.
* Patient has a history of or known esophageal stricture or gross esophageal anatomic abnormalities (Schatzki's ring, obstructive lesions, etc.).
* Patient has esophageal or gastric varices.
* Patient has Barrett's esophagus.
* Patient cannot understand trial requirements or is unable to comply with follow-up schedule.
* Pregnant or nursing, or plans to become pregnant during the course of the study.
* Any reason which the Investigator believes may cause the subject to be non-compliant with or unable to meet the protocol requirements.
* Patient has an electrical implant or metallic, abdominal implants.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change is GERD-HRQL Score as a measure of efficacy | Baseline, 6 month visit
Number of participants with serious complications as a measure of safety. | 6 month visit
Change is total distal acid exposure as a measure of efficacy. | Baseline, 6 month visit

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (3):
  - Schön Klinik Nürnberg, Fürth
  - EvK Herne, Herne
  - Uni Klinik Leipzig, Leipzig
- Policlinico San Donato, Milan, Italy